CLINICAL TRIAL: NCT04347005
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Rising Dose Study of AR882, a Potent Uricosuric Agent, in Healthy Adult Male Volunteers
Brief Title: The Study is Designed to Evaluate Single Ascending Doses of AR882 in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arthrosi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR882-101
Record Dates: First submitted 2020-03-10; First posted 2020-04-15 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Allopurinol; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- AR882 (Dose A) (Experimental)
  Interventions: Drug: Cohort 1: AR882
- AR882 (Dose B) (Experimental)
  Interventions: Drug: Cohort 2: AR882; Drug: Cohort 6: AR882 Food Effect; Drug: Cohort 8: AR882 in combination with allopurinol; Drug: Cohort 9: AR882 in combination with febuxostat
- AR882 (Dose C) (Experimental)
  Interventions: Drug: Cohort 3: AR882
- AR882 (Dose D) (Experimental)
  Interventions: Drug: Cohort 4: AR882
- AR882 (Dose E) (Experimental)
  Interventions: Drug: Cohort 5: AR882
- AR882 (Dose B) Solid Oral Formulation (Experimental)
  Interventions: Drug: Cohort 7: AR882 Solid Oral Formulation
- Placebo (Placebo Comparator)
  Interventions: Drug: Cohort 1: AR882; Drug: Cohort 2: AR882; Drug: Cohort 3: AR882; Drug: Cohort 4: AR882; Drug: Cohort 5: AR882; Drug: Cohort 6: AR882 Food Effect; Drug: Cohort 7: AR882 Solid Oral Formulation
- Allopurinol (Active Comparator)
  Interventions: Drug: Cohort 8: AR882 in combination with allopurinol
- Febuxostat (Active Comparator)
  Interventions: Drug: Cohort 9: AR882 in combination with febuxostat

INTERVENTIONS:
Drug: Cohort 1: AR882 — Single dose of AR882 or matching placebo
  Arms: AR882 (Dose A); Placebo
Drug: Cohort 2: AR882 — Single dose of AR882 or matching placebo
  Arms: AR882 (Dose B); Placebo
Drug: Cohort 3: AR882 — Single dose of AR882 or matching placebo
  Arms: AR882 (Dose C); Placebo
Drug: Cohort 4: AR882 — Single dose of AR882 or matching placebo
  Arms: AR882 (Dose D); Placebo
Drug: Cohort 5: AR882 — Single dose of AR882 or matching placebo
  Arms: AR882 (Dose E); Placebo
Drug: Cohort 6: AR882 Food Effect — Single dose of AR882 or matching placebo in a fed state
  Arms: AR882 (Dose B); Placebo
Drug: Cohort 7: AR882 Solid Oral Formulation — Single dose of AR882 or matching placebo
  Arms: AR882 (Dose B) Solid Oral Formulation; Placebo
Drug: Cohort 8: AR882 in combination with allopurinol — Single dose of allopurinol alone and a single dose of AR882 in combination with a single dose of allopurinol
  Arms: AR882 (Dose B); Allopurinol
Drug: Cohort 9: AR882 in combination with febuxostat — Single dose of febuxostat alone and a single dose of AR882 in combination with a single dose of febuxostat
  Arms: AR882 (Dose B); Febuxostat

SUMMARY:
A randomized, double-blind, placebo-controlled, single ascending dose study of AR882 in healthy adult males.

ELIGIBILITY:
Inclusion Criteria:

* Serum uric acid level ≥ 4.5 mg/dL (268 µmol/L)
* Body weight no less than 50 kg and body mass index (BMI) within the range of ≥18 and ≤33 kg/m2
* Must be free of any clinically significant disease that requires a physician's care and/or would interfere with study evaluations or procedures

Exclusion Criteria:

* Malignancy within 5 years, except for successfully treated basal or squamous cell carcinoma of the skin
* History of cardiac abnormalities
* History and/or presence of drug addiction or excessive use of alcohol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety profile of AR882 based on incidence of abnormal laboratory findings | 8 Days
  Analysis of abnormal safety laboratory findings
Safety Analyses | 8 Days
  ECG Heart Rate
Safety Analyses | 8 Days
  ECG PR-Interval
Safety Analyses | 8 Days
  ECG RR-Interval
Safety Analyses | 8 Days
  ECG QRS-Interval
Safety Analyses | 8 Days
  ECG QT-Interval
Safety Analyses | 8 Days
  ECG QTc-Interval
Safety Analyses | 8 Days
  Vital Sign - Systolic Blood Pressure
Safety Analyses | 8 Days
  Vital Sign - Diastolic Blood Pressure
Safety Analyses | 8 Days
  Vital Sign - Pulse Rate
Safety Analyses | 8 Days
  Vital Sign - Body Temperature
Safety Analyses | 8 Days
  Vital Sign - Respiratory Rate
Area under the curve (AUC) for plasma AR882 | 6 Days
  Profile from plasma in terms of AUC for AR882
Time to maximum plasma concentration (Tmax) for AR882 | 6 Days
  Profile from plasma in terms of Tmax for AR882
Maximum plasma concentration (Cmax) for AR882 | 6 Days
  Profile from plasma in terms of Cmax for AR882
Apparent terminal half-life (t1/2) for AR882 | 6 Days
  Profile from plasma in terms of t1/2 for AR882
Amount excreted (Ae) into urine for AR882 | 6 Days
  Profile from urine in terms of Ae for AR882
Fractional Excretion (FEUA) for AR882 | 6 Days
  Profile from urine in terms of FEUA for AR882

SECONDARY OUTCOMES:
PD profile of a single dose of AR882 | 6 Days
  Profile from serum uric acid concentrations over time
PD profile of a single dose of AR882 in combination with allopurinol | 6 Days
  Profile from serum uric acid concentrations over time
PD profile of a single dose of AR882 in combination with febuxostat | 6 Days
  Profile from serum uric acid concentrations over time

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty, Ltd., Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No